CLINICAL TRIAL: NCT00922675
Title: Postconditioning in ST-elevation Myocardial Infarction Treated With Primary PCI
Brief Title: Postconditioning in ST-elevation Myocardial Infarction
Acronym: POSTEMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Jan Eritsland, Senior Consultant Cardiology, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Po 1506
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Myocardial Infarction
Keywords: ST-elevation myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — Ischemic Postconditioning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Postconditioning (Experimental): Active arm:Postconditioning protocol before routine PCI/stenting of an occluded coronary artery
  Interventions: Procedure: Postconditioning
- Control (Other): Control arm: Routine PCI/stenting of an occluded coronary artery without postconditioning
  Interventions: Procedure: Control intervention

INTERVENTIONS:
Procedure: Postconditioning — After opening of IRA and establishment of TIMI-flow grade 2 or 3, the control group continues the procedure with stenting. In the postconditioning group 4 additional balloon inflations separated by 1 minute reperfusion are given, starting after 1 minute of reperfusion.
  Arms: Postconditioning
Procedure: Control intervention — After opening of IRA and establishment of TIMI-flow grade 2 or 3, the control group continues the procedure with stenting.
  Arms: Control

SUMMARY:
Study objectives: To assess the effects of postconditioning on infarct size in patients with ST-elevation infarction referred to PCI.

Study design: Prospective, randomized, open-label study with blinded endpoint evaluation. Included patients will be randomly allocated to postconditioning or control. Patients with symptoms of acute myocardial infarction of less than 6 hours duration fulfilling ECG criteria for primary PCI are eligible. PCI follow established routines. In postconditioning patients, additional, short (1 min), intermittent balloon occlusions will be applied after initial opening of infarct related artery. After this intervention, PCI proceeds routinely with stent implantation. In the control group, stent implantation after initial opening proceeds as usual. Primary endpoint is final infarct size, determined by MRI after 4 months. 260 patients will be included. Follow-up is 1 year. Inclusion period: 18 - 24 months.

Clinical implications: Reperfusion therapy, administered as early as possible after start of symptoms, has improved the prognosis in acute ST-elevation myocardial infarction. Still, however, many patients suffer large infarctions, subsequently with an increased risk of heart failure, arrhythmias, and death. In pilot studies, mechanical postconditioning has been shown to reduce infarct size and thus potentially improve prognosis. However, the effect of postconditioning must be confirmed in larger clinical trials before implemented in routine treatment.

ELIGIBILITY:
Inclusion Criteria:

* acute symptoms consistent with an acute myocardial infarction of less than 6 hours duration
* an occluded infarct related artery must be demonstrated (TIMI-flow 0-1)

Exclusion Criteria:

* Prior myocardial infarction
* Demonstration of collaterals to the infarcted area
* TIMI-flow >1 before intervention or TIMI-flow <2 after initial balloon inflation
* Demonstration of a distal occlusion
* Patients given thrombolytic treatment
* Patients in cardiogenic shock
* Any contraindication to MRI (magnetic resonance imaging)
* Unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2009-06; Primary Completion 2012-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Infarct size, assessed by MRI | 4 months

SECONDARY OUTCOMES:
Myocardial blushing grade | assessed at the end of PCI procedure
ST-resolution in ECG | Assessed after 1 hour
Troponin-T and CK-MB | peak release values
Echocardiographic evaluation of left ventricular function including speckle-tracking measurement. | assessed at baseline, 4 months and1 year
  Assesment of LV function. Comparison with CMR in the whole study population and between treatment groups.
Incidence of treated arrhythmias and heart failure during initial hospitalization Incidence of death, non-fatal myocardial infarction, unstable angina, heart failure, and cerebrovascular disease | 1-year follow up.
Myocardial salvage | Baseline to 4 months
  Myocardial salvage defined as (area at risk-final infarct size)/area at risk. Area at risk measured by CMR at baseline and final infarct size by CMR at 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Eritsland, MD, PhD, Study Chair — Oslo Univ.Hosp. Ulleval
Locations (1):
- Dept. of Cardiology, Oslo Univ. Hosp. Ulleval, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tollefsen IM, Shetelig C, Seljeflot I, Eritsland J, Hoffmann P, Andersen GO. High levels of interleukin-6 are associated with final infarct size and adverse clinical events in patients with STEMI. Open Heart. 2021 Dec;8(2):e001869. doi: 10.1136/openhrt-2021-001869. PMID 34933964
- [Derived] Limalanathan S, Andersen GO, Klow NE, Abdelnoor M, Hoffmann P, Eritsland J. Effect of ischemic postconditioning on infarct size in patients with ST-elevation myocardial infarction treated by primary PCI results of the POSTEMI (POstconditioning in ST-Elevation Myocardial Infarction) randomized trial. J Am Heart Assoc. 2014 Apr 23;3(2):e000679. doi: 10.1161/JAHA.113.000679. PMID 24760962